CLINICAL TRIAL: NCT00528177
Title: Phase 4: A Comparison of Intravenous Administration of Morphine vs. Oxycodone for Postoperative Pain Management Following Laparoscopic Hysterectomy or Myomectomy
Brief Title: Morphine vs. Oxycodone for Postoperative Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Ullevaal University Hospital, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 328-07137 1.2007.1463
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-06

CONDITIONS: Hysterectomy; Myoma; Postoperative Pain; Opioids
Keywords: kappa-opioid receptor; my-opioid receptor; oxycodone; morphine; postoperative pain
MeSH Terms: conditions — Myoma; Pain, Postoperative | interventions — MoxDuo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- O (Active Comparator): This arm will receive intravenous oxycodone at the end of surgery and PCA oxycodone for postoperative pain relief.
  Interventions: Drug: Morphine and oxycodone
- M (Active Comparator): This arm will receive intravenous morphine at the end of surgery and PCA morphine for postoperative pain relief.
  Interventions: Drug: Morphine and oxycodone

INTERVENTIONS:
Drug: Morphine and oxycodone — At the end of surgery, group 1 will receive intravenous morphine 0.07 mg/kg and intravenous PCA morphine 0.015 mg/kg every time they push the botton with 5 minutes lock-out interval. Maximum 16 mg/2 hours. Group 2 will receive intravenous oxycodone 0.07 mg/kg and intravenous PCA oxycodone 0.015 mg/kg every time they push the botton with 5 minutes lock-out interval. Maximum 16 mg/2 hours.
  The patients will use the PCA until the next morning.

SUMMARY:
The purpose of this study is to determine whether oxycodone provides better analgesia compared to morphine after laparoscopic hysterectomy or myomectomy.

DETAILED DESCRIPTION:
Traditionally, a 1:1 ratio in analgesic potency between intravenous morphine and oxycodone has been presumed (1-2), but one study demonstrated a 3:2 ratio between those drugs (3). During the last years, several studies indicate that oxycodone has the potential of mediating pain relief through the kappa-opioid receptor (4-6), and not only on the my-opioid receptor like most other opioids used in the clinic. Kappa-opioid receptors are widely distributed in visceral organs, and this may explain why Kalso (3) found less need for oxycodone compared to morphine in patients undergoing abdominal surgery.

The aim of this study is to investigate whether patients with visceral postoperative pain need less oxycodone compared to morphine, and whether patients receiving oxycodone experience better pain relief and less adverse effects compared to patients receiving morphine.

Before start of surgery, the patients will be tested with PainMatcher, an instrument testing electrical pain threshold in the skin (7-10), to ensure that both groups have the same pain threshold before surgery.

References

1. Kalso E. Oxycodone. Journal of Pain & Symptom Management 2005; 29: S47-S56.
2. Silvasti M, Rosenberg P, Seppala T, Svartling N, Pitkanen M. Comparison of analgesic efficacy of oxycodone and morphine in postoperative intravenous patient-controlled analgesia. Acta Anaesthesiol Scand 1998; 42: 576-80.
3. Kalso E, Poyhia R, Onnela P, Linko K, Tigerstedt I, Tammisto T. Intravenous morphine and oxycodone for pain after abdominal surgery. Acta Anaesthesiol Scand 1991; 35: 642-6.
4. Staahl C, Christrup LL, Andersen SD, Arendt-Nielsen L, Drewes AM. A comparative study of oxycodone and morphine in a multi-modal, tissue-differentiated experimental pain model. Pain 2006; 123: 28-36.
5. Ross FB, Smith MT. The intrinsic antinociceptive effects of oxycodone appear to be kappa-opioid receptor mediated. Pain 1997; 73: 151-7.
6. Sandner-Kiesling A, Pan HL, Chen SR, James RL, Haven-Hudkins DL, Dewan DM, Eisenach JC. Effect of kappa opioid agonists on visceral nociception induced by uterine cervical distension in rats. Pain 2002; 96: 13-22.
7. Alstergren P, Forstrom J, Alstergren P, Forstrom J. Acute oral pain intensity and pain threshold assessed by intensity matching to pain induced by electrical stimuli. Journal of Orofacial Pain 2003; 17: 151-9.
8. Lundeberg T, Lund I, Dahlin L, Borg E, Gustafsson C, Sandin L, Rosen A, Kowalski J, Eriksson SV. Reliability and responsiveness of three different pain assessments. Journal of Rehabilitation Medicine 2001; 33: 279-83.
9. Nielsen PR. Prediction of post-operative pain by an electrical pain stimulus. Acta Anaesthesiol Scand 2007; 51: 582-6.
10. Stener-Victorin E, Kowalski J, Lundeberg T. A new highly reliable instrument for the assessment of pre- and postoperative gynecological pain. Anesth & Analg 95: 151-7.

ELIGIBILITY:
Inclusion Criteria:

* Patients (American Society of Anaesthesiologists (ASA) I, II and III) due for elective, laparoscopic, non-malignant gynaecologic surgery: Hysterectomy or myomectomy.
* Written informed consent.
* Age: 18 to 70 years.

Exclusion Criteria:

* Patients having used non-steroidal anti-inflammatory drugs (NSAIDs) the last 24 hours.
* Sensitivity towards the study drugs.
* Cardiovascular risk conditions: Heart failure, unstable hypertension, coronary artery disease.
* Patients using opioids, steroids or anti-emetic drugs.
* Serious mental disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Dosage relation between oxycodone and morphine. Pain score (VAS). Adverse effects. | Within the first postoperative day (24 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Johan Ræder, Prof.MD,Phd, Study Director — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Lenz H, Sandvik L, Qvigstad E, Bjerkelund CE, Raeder J. A comparison of intravenous oxycodone and intravenous morphine in patient-controlled postoperative analgesia after laparoscopic hysterectomy. Anesth Analg. 2009 Oct;109(4):1279-83. doi: 10.1213/ane.0b013e3181b0f0bb. PMID 19762758